CLINICAL TRIAL: NCT07337928
Title: Altitude Training Effectiveness; Is There a Role for Sleep and Menstrual Health?
Acronym: FEMHEALTH
Status: Not yet recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Royal Military Academy (Unknown)
Responsible Party: Principal Investigator, Bart Roelands, Professor, Vrije Universiteit Brussel
Other Study IDs: FEMHEALTH
Record Dates: First submitted 2025-11-28; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Altitude Effectiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite female cyclists: Elite female cyclists participating in an altitude training camp

SUMMARY:
Therefore, the present study aims to evaluate the role of the impact of altitude on sleep and the menstrual cycle in the inter- and intraindividual variability of altitude training effectiveness. In order to do so, elite female cyclists will be monitored before, during and after an altitude training camp. The monitoring will include menstrual cycle characteristics, sleep and altitude effectiveness and will start three months before the start of the altitude training camp and end two months after the altitude training camp. Both naturally cycling women and women using contraceptives will be included in the study. Menstrual cycle monitoring will take place via self-reports and via a daily saliva (Eli Health) and urine (Proov) test to measure progesterone concentration. Besides proges-terone concentration, the sampled urine will also be used to perform an ovulation test on (i.e., measuring the luteinizing hormone). In addition, a blood sample will be collected at the start of each menstrual cycle to evaluate the concentration of menstrual cycle-related hormones (e.g., fol-licle-stimulating hormone, luteinizing hormone, estrogen, and progesterone) and to evaluate the functioning of the Hypothalamic-Pituitary-Adrenal Axis (i.e., cortisol concentration). Sleep moni-toring will be performed via the use of questionnaires, actigraphy and polysomnography. Lastly, altitude effectiveness will be evaluated via the altitude-associated response in total hemoglobin mass and via an all out cycle ergometer task.

DETAILED DESCRIPTION:
Elite athletes are constantly aiming to improve their performance and, eventually, outperform their opponents. In this endeavor, various methods have been designed to gain an advantage over the other competitors. One of those methods, which has been in use for quite some time and remains very popular, is altitude training. Currently, multiple protocols of altitude training have been developed. A general distinction can be made between "live high, train high" (LHTH), "live high, train low" (LHTL), and "live low, train high" (LLTH) altitude training. The LHTL protocol is cur-rently being put forward as the most effective one for training gains.

The overall effectiveness of altitude training to improve performance is backed up by a significant amount of scientific data. Nonetheless, up to date, the efficacy of altitude training is still questioned by some, due the lack of rigorous and well-controlled investigations, and no scientific consensus exists. Since Lundby and colleagues published their critical views on the general application of altitude training to enhance performance in elite athletes, follow-up research has substantiated these critical views of Lundby and colleagues. Nevertheless, the debate on the usefulness of altitude training in elite athletes is still ongoing, and currently revolves around whether athletes with an already high hemoglobin mass (i.e., elite athletes) can successfully increase their hemoglobin mass via altitude training.

A topic that could provide some new insights is the issue of intra- and interindividual variability in the response to altitude training, and the underlying mechanisms of these variabilities. Multiple studies have been performed that clearly outline the presence of both intra- and interindividual variability in the response to altitude training. The determination and evaluation of all state and trait-specific factors that could influence an athlete's response to altitude training is cur-rently ongoing. Nummela et al. showed that the mean effectiveness of altitude training in yielding an increase in hemoglobin mass could rise from 56% to 69% when targeting altitude exposure (2,000-2,500 m), iron deficiency and inflammation as moderating state factors. This emphasizes the need to carefully consider all the possible moderating state factors that may influence an athlete's response to altitude training. Furthermore, these findings stress the need for future research to describe more accurately how these different influencing state factors (and potential oth-er state and trait factors) interact to impact the altitude training-response in both elite and recrea-tional athletes.

One of these potentially crucial factors that could play a role in the effectiveness of altitude training to trigger performance-improving adaptations is sleep. Sleep is one of the most important aspects of recovery, and nowadays it is recommended to stay below 3,000 m (or an equivalent normobaric reduction of inspired O2) at night in altitude training paradigms. This recommendation is based on the fact that sleep is impaired at high altitude, and impaired sleep could counteract the positive physiological responses that are aimed for, certainly when it is prolonged for ~2-3 weeks (i.e., the current suggested optimal hypoxic dose, taking into account altitude and exposure time [1]). However, the guideline to stay below 3,000 m to prevent altitude-induced sleep impairments might be inadequate. Hoshikawa et al. demonstrated that acute exposure to normobaric hypoxia equivalent to a 2,000 m altitude decreased slow-wave sleep in athletes, but it did not change subjective sleepiness or amounts of urinary catecholamines. These results point out that the athlete's sleep might be disturbed even at moderate altitudes of 2,000 m and, more importantly, that athletes are not aware of it (i.e., subjective sleepiness did not change). Moreover, the study of Hoshikawa et al. also revealed that the apnea/hypopnea index (AHI; i.e., the number of signif-icant respiratory events qualifying as apnea or hypopnea per hour of sleep) increased in hypoxia compared to normoxia, and the magnitude of this effect varied widely among participants (i.e., high interindividual variability). This high interindividual variability might be associated with the interindividual variability that is observed in altitude training effectiveness. A hypothesis that is further substantiated by the recently published data of Mujika et al., that demonstrates a link between subjective sleep quality and the effectiveness of altitude training to increase total hemo-globin mass.

Specifically within female athletes, another potential crucial factor in the effectiveness of altitude training is the hypothalamic-pituitary-ovarian (HPO) axis function. The hypothalamic-pituitary-ovarian (HPO) axis regulates reproductive function, including the orchestration of ovula-tion and menstrual cyclicity. HPO axis suppression leads to altered hormonal patterns and conse-quently short luteal phases, anovulation and amenorrhoea. Shaw et al. concluded in their sys-tematic review that, if lowlanders travel to highland for short or longer duration, the high altitude-hypoxia affects their menstrual cycle more adversely than the natives. The variation in female hormones may contribute in unsuccessful ovulation, menstrual cycle, and subsequently pregnancy at high altitude. A disturbed HPO axis function at altitude can, subsequently, negatively im-pact the effectiveness of altitude training. For example, Heikura et al. recently reported lower pre-hypoxic exposure hemoglobin mass levels in amenorrheic versus eumenorrheic women, sug-gesting that menstrual dysfunction, an indicator of long-term low energy availability, may influence the altitude exposure-related increase in hemoglobin mass or its magnitude.

Therefore, the present study aims to evaluate the role of the impact of altitude on sleep and the menstrual cycle in the inter- and intraindividual variability of altitude training effectiveness. In order to do so, elite female cyclists will be monitored before, during and after an altitude training camp. The monitoring will include menstrual cycle characteristics, sleep and altitude effectiveness and will start three months before the start of the altitude training camp and end two months after the altitude training camp. Both naturally cycling women and women using contraceptives will be included in the study. Menstrual cycle monitoring will take place via self-reports and via a daily saliva (Eli Health) and urine (Proov) test to measure progesterone concentration. Besides proges-terone concentration, the sampled urine will also be used to perform an ovulation test on (i.e., measuring the luteinizing hormone). In addition, a blood sample will be collected at the start of each menstrual cycle to evaluate the concentration of menstrual cycle-related hormones (e.g., follicle-stimulating hormone, luteinizing hormone, estrogen, and progesterone) and to evaluate the functioning of the Hypothalamic-Pituitary-Adrenal Axis (i.e., cortisol concentration). Sleep monitoring will be performed via the use of questionnaires, actigraphy and polysomnography. Lastly, altitude effectiveness will be evaluated via the altitude-associated response in total hemoglobin mass and via an all out cycle ergometer task.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female
* Elite cyclist

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligibility criteria are being a healthy female elite cyclist. Both naturally cycling women and women who use contraception are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Total hemoglobin mass (tHBmass) | Will be measured at sea level 5 days before (i.e., Day -5) and on the last day of the altitude training camp (i.e., Day 18)
  An optimized carbon monoxide rebreathing method will be used. The carbon monoxide dose will be 0.8 mL/kg body mass. The rebreathing procedure will be performed for 2 minutes, in a seated position, through a glass spirometer.
A standardized 5-min all-out cycling test | Will be performed on a calibrated cycle ergometer 5 days before (i.e. Day -5) and on the final day of the altitude training camp (i.e., Day 18)
  After a 10-15 min warm-up, participants will complete a maximal 5-min effort in linear (cadence-dependent) mode, during which they will be instructed to produce the highest sustainable power for the entire duration. Power output, cadence, and heart rate will be recorded continuously. Mean 5-min power (W and W·kg-¹) will serve as the primary performance outcome, with peak power and end-segment power examined as secondary metrics.
A wake and sleep diary | Participants will have to fill out this wake and sleep diary daily from Day -7 to Day 25 (Day 0 being the first day of the altitude training camp).
  Will be used regarding sleep (completed by participants the morning upon waking) and daytime activity (completed prior to their bedtime). The participants have to indicate, on a 24-h scale with a time resolution of 15 min, 1) when they started trying to fall asleep, 2) when they actually fell asleep, 3) whether they woke up after falling asleep and, if yes, for how long, 4) when they woke up, and 5) whether they took a nap out of bed and, if yes, for how long. Subsequently, the following outcome measures will be calculated: total time spent in bed, sleep onset latency, wake after sleep onset, total sleep time, total nap time, bed-time and risetime. In addition, participants will also be asked to rate their sleep quality, quality of the wake-up and shape of the day (score on a 10-point scale).
The Pittsburgh Sleep Quality Index (PSQI) | The PSQI will have to be completed at the end of each month in which the menstrual cyclus is monitored (i.e., Month -3 final day, Month -2 final day, Month -1 final day, Month 0 final day, Month 1 final day and Month 2 final day).
  The PSQI includes 19 self-assessment items that combine to give 7 components of the overall score, with each component receiving a score of 0 to 3. A score of 0 indicates no difficulty, while a score of 3 indicates severe difficulty. The 7 components of the score add up to give an overall score ranging from 0 to 21 points, with 0 indicating no difficulty and 21 indicating major difficul-ties. An overall sum of 5 or more indicates a 'bad' sleeper.
Actigraphy | The participants will be requested to wear the ActiGraph for a period of 24 hours without interruption on Day -7, Day -6, Day 0, Day 1, Day 6, Day 7, Day 12, Day 13, Day 17, Day 18, Day 24 en Day 25 (Day 0 being the start of the altitude training camp).
  Sleep measures will be assessed by non-dominant wrist-worn actigraphy with the ActiGraph wGT3X-BT device from Ametris and data will be collected with a sampling frequency of 30-50hz. The ActiGraph output variables will be total sleep time (TST, in min), total time in bed (TTB, in min), sleep onset latency (SOL, in min), wake after sleep onset (WASO, in min), number of awak-ening after sleep onset (nAw, number) and sleep efficiency (SE in %, the ratio between total sleep time and total time spent in bed) in agreement with the guidelines of the Society of Behavioral Sleep Medicine.
Polysomnography | Will be used to monitor sleep on pre Day -7, Day -7, Day 1, Day 6, Day 12, Day 18 en Day 25 (Day 0 being the start of altitude training camp).
  The SomnoTouch RESP system (SomnoMedics GmbH, Germany), a portable, Type III sleep diagnostic device will be used to perform ambulatory polysomnography. The device records respiratory effort, nasal airflow, blood oxygen saturation, heart rate, actigraphy, body position, and bilateral thoracic bio-impedance signals. Data will be collected in accordance with manufacturer specifications and validated scoring standards.
A survey which documents menstrual cycle history | Once, at the start of the monitoring period, 3 months prior the altitude training camp.
  Any current or previous hormonal contraception use (type, formulation), the length and frequency of their menstrual cycle (including determination of any primary and secondary amenorrhea) and prevalence of known menstrual diagnoses (e.g., polycystic ovary syndrome [PCOS], endometriosis) will be documented.
A short questionnaire asking whether they bled, flow and cramping. | On a daily basis. This daily basis monitoring will start three months before the start of the altitude training camp, and will end two months after the altitude training camp.
  A short questionnaire asking whether they bled (+ form of bleeding; withdrawal, breakthrough or spotting bleeding), flow (light/medium/heavy) and cramping (0-10).
A saliva (Eli Health) test | This daily testing will start 3 months before the start of the altitude training camp and end two months after the altitude training camp.
  To measure progesterone concentration
A urine (Proov) test | This daily testing will start 3 months before the start of the altitude training camp and end two months after the altitude training camp.
  To measure progesterone concentration
A urine sample | The ovulation test will have to be performed starting several days before the expected luteinizing hormone surge so that the peak is not missed (i.e., Day 7 of the cycle) and stop on Day 18 of the cycle (each cycle is 28 days).
  To perform an ovulation test on (i.e., measuring the luteinizing hormone).
A blood sample | At the start of each menstrual cycle during the monitoring period (from three months before the altitude training camp till two months after the altitude training camp).
  To evaluate the concentration of menstrual cycle-related hormones (e.g., follicle-stimulating hormone, luteinizing hormone, estrogen, and progesterone) and to evaluate the functioning of the Hy-pothalamic-Pituitary-Adrenal Axis (i.e., cortisol concentration).

IPD SHARING:
Plan to Share IPD: No
Given that we will be working with elite cyclists, the IPD will be confidential.

REFERENCES:
- [Background] Heikura IA, Burke LM, Bergland D, Uusitalo ALT, Mero AA, Stellingwerff T. Impact of Energy Availability, Health, and Sex on Hemoglobin-Mass Responses Following Live-High-Train-High Altitude Training in Elite Female and Male Distance Athletes. Int J Sports Physiol Perform. 2018 Sep 1;13(8):1090-1096. doi: 10.1123/ijspp.2017-0547. Epub 2018 Sep 13. PMID 29431548
- [Background] Shaw S, Ghosh D, Kumar U, Panjwani U, Kumar B. Impact of high altitude on key determinants of female reproductive health: a review. Int J Biometeorol. 2018 Nov;62(11):2045-2055. doi: 10.1007/s00484-018-1609-0. Epub 2018 Sep 14. PMID 30218203
- [Background] Burtscher J, Raberin A, Brocherie F, Malatesta D, Manferdelli G, Citherlet T, Krumm B, Bourdillon N, Antero J, Rasica L, Burtscher M, Millet GP. Recommendations for Women in Mountain Sports and Hypoxia Training/Conditioning. Sports Med. 2024 Apr;54(4):795-811. doi: 10.1007/s40279-023-01970-6. Epub 2023 Dec 12. PMID 38082199
- [Background] Mujika I, Tian R, Zelenkova I, Pyne DB. Highly Variable Hemoglobin-Mass Changes During Successive Altitude Training Camps in World-Class Female Water Polo Players. Int J Sports Physiol Perform. 2025 Oct 28;20(12):1763-1767. doi: 10.1123/ijspp.2025-0270. Print 2025 Dec 1. PMID 41151548
- [Background] Hoshikawa M, Uchida S, Sugo T, Kumai Y, Hanai Y, Kawahara T. Changes in sleep quality of athletes under normobaric hypoxia equivalent to 2,000-m altitude: a polysomnographic study. J Appl Physiol (1985). 2007 Dec;103(6):2005-11. doi: 10.1152/japplphysiol.00315.2007. Epub 2007 Aug 9. PMID 17690200
- [Background] West, J.B., et al., Sleep, in High altitude medicine and physiology, J.B.S. West, Robert B, A.M. Luks, and J.S. Milledge, Editors. 2013, CRC Press: Padstow, Cornwall.
- [Background] McLean BD, Buttifant D, Gore CJ, White K, Liess C, Kemp J. Physiological and performance responses to a preseason altitude-training camp in elite team-sport athletes. Int J Sports Physiol Perform. 2013 Jul;8(4):391-9. doi: 10.1123/ijspp.8.4.391. Epub 2012 Nov 19. PMID 23170749
- [Background] McLean BD, Buttifant D, Gore CJ, White K, Kemp J. Year-to-year variability in haemoglobin mass response to two altitude training camps. Br J Sports Med. 2013 Dec;47 Suppl 1(Suppl 1):i51-8. doi: 10.1136/bjsports-2013-092744. PMID 24282208
- [Background] Hauser A, Troesch S, Saugy JJ, Schmitt L, Cejuela-Anta R, Faiss R, Steiner T, Robinson N, Millet GP, Wehrlin JP. Individual hemoglobin mass response to normobaric and hypobaric "live high-train low": A one-year crossover study. J Appl Physiol (1985). 2017 Aug 1;123(2):387-393. doi: 10.1152/japplphysiol.00932.2016. Epub 2017 May 18. PMID 28522767
- [Background] Friedmann B, Frese F, Menold E, Kauper F, Jost J, Bartsch P. Individual variation in the erythropoietic response to altitude training in elite junior swimmers. Br J Sports Med. 2005 Mar;39(3):148-53. doi: 10.1136/bjsm.2003.011387. PMID 15728692
- [Background] Chapman RF, Stray-Gundersen J, Levine BD. Individual variation in response to altitude training. J Appl Physiol (1985). 1998 Oct;85(4):1448-56. doi: 10.1152/jappl.1998.85.4.1448. PMID 9760340
- [Background] Millet GP, Chapman RF, Girard O, Brocherie F. Is live high-train low altitude training relevant for elite athletes? Flawed analysis from inaccurate data. Br J Sports Med. 2019 Aug;53(15):923-925. doi: 10.1136/bjsports-2017-098083. Epub 2017 Dec 15. No abstract available. PMID 29247024
- [Background] Racinais S, Periard JD, Piscione J, Bourdon PC, Cocking S, Ihsan M, Lacome M, Nichols D, Townsend N, Travers G, Wilson MG, Girard O. Intensified Training Supersedes the Impact of Heat and/or Altitude for Increasing Performance in Elite Rugby Union Players. Int J Sports Physiol Perform. 2021 Mar 5;16(10):1416-1423. doi: 10.1123/ijspp.2020-0630. Epub 2021 Mar 5. PMID 33668015
- [Background] Bejder J, Andersen AB, Buchardt R, Larsson TH, Olsen NV, Nordsborg NB. Endurance, aerobic high-intensity, and repeated sprint cycling performance is unaffected by normobaric "Live High-Train Low": a double-blind placebo-controlled cross-over study. Eur J Appl Physiol. 2017 May;117(5):979-988. doi: 10.1007/s00421-017-3586-0. Epub 2017 Mar 22. PMID 28332025
- [Background] Robach P, Hansen J, Pichon A, Meinild Lundby AK, Dandanell S, Slettalokken Falch G, Hammarstrom D, Pesta DH, Siebenmann C, Keiser S, Kerivel P, Whist JE, Ronnestad BR, Lundby C. Hypobaric live high-train low does not improve aerobic performance more than live low-train low in cross-country skiers. Scand J Med Sci Sports. 2018 Jun;28(6):1636-1652. doi: 10.1111/sms.13075. Epub 2018 Mar 22. PMID 29469995
- [Background] Bejder J, Nordsborg NB. Specificity of "Live High-Train Low" Altitude Training on Exercise Performance. Exerc Sport Sci Rev. 2018 Apr;46(2):129-136. doi: 10.1249/JES.0000000000000144. PMID 29346162
- [Background] Lundby C, Robach P. Does 'altitude training' increase exercise performance in elite athletes? Exp Physiol. 2016 Jul 1;101(7):783-8. doi: 10.1113/EP085579. Epub 2016 Jun 13. PMID 27173805
- [Background] Lundby C, Millet GP, Calbet JA, Bartsch P, Subudhi AW. Does 'altitude training' increase exercise performance in elite athletes? Br J Sports Med. 2012 Sep;46(11):792-5. doi: 10.1136/bjsports-2012-091231. Epub 2012 Jul 14. PMID 22797528
- [Background] Gore CJ, Sharpe K, Garvican-Lewis LA, Saunders PU, Humberstone CE, Robertson EY, Wachsmuth NB, Clark SA, McLean BD, Friedmann-Bette B, Neya M, Pottgiesser T, Schumacher YO, Schmidt WF. Altitude training and haemoglobin mass from the optimised carbon monoxide rebreathing method determined by a meta-analysis. Br J Sports Med. 2013 Dec;47 Suppl 1(Suppl 1):i31-9. doi: 10.1136/bjsports-2013-092840. PMID 24282204
- [Background] Wilber RL. Current trends in altitude training. Sports Med. 2001;31(4):249-65. doi: 10.2165/00007256-200131040-00002. PMID 11310547
- [Background] Mujika I, Sharma AP, Stellingwerff T. Contemporary Periodization of Altitude Training for Elite Endurance Athletes: A Narrative Review. Sports Med. 2019 Nov;49(11):1651-1669. doi: 10.1007/s40279-019-01165-y. PMID 31452130
- [Background] Bonetti DL, Hopkins WG. Sea-level exercise performance following adaptation to hypoxia: a meta-analysis. Sports Med. 2009;39(2):107-27. doi: 10.2165/00007256-200939020-00002. PMID 19203133
- [Background] Billaut F, Gore CJ, Aughey RJ. Enhancing team-sport athlete performance: is altitude training relevant? Sports Med. 2012 Sep 1;42(9):751-67. doi: 10.1007/BF03262293. PMID 22845561
- [Background] Girard O, Amann M, Aughey R, Billaut F, Bishop DJ, Bourdon P, Buchheit M, Chapman R, D'Hooghe M, Garvican-Lewis LA, Gore CJ, Millet GP, Roach GD, Sargent C, Saunders PU, Schmidt W, Schumacher YO. Position statement--altitude training for improving team-sport players' performance: current knowledge and unresolved issues. Br J Sports Med. 2013 Dec;47 Suppl 1(Suppl 1):i8-16. doi: 10.1136/bjsports-2013-093109. PMID 24282213
- [Background] Nummela A, Eronen T, Koponen A, Tikkanen H, Peltonen JE. Variability in hemoglobin mass response to altitude training camps. Scand J Med Sci Sports. 2021 Jan;31(1):44-51. doi: 10.1111/sms.13804. Epub 2020 Sep 9. PMID 32783231